CLINICAL TRIAL: NCT03836456
Title: Defining Approaches That Support the Mental Health of Post-secondary Students Who Experienced More Than Three Adverse Childhood Experiences
Brief Title: Approaches That Support Mental Health in Post-secondary Students With Adverse Childhood Experiences
Acronym: ACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Rob Gilbert, Associate Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DalhousieU
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Adverse Childhood Experiences; Mindfulness; Students

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data collected will be coded and codes will not be revealed to the investigators or outcome assessors until after data analysis is complete. The study participants will be told they are participating in an intervention to promote mental health but not told which of the 2 interventions is the active control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention (Experimental): Mindfulness Based Stress Resilience Training: This approach will be conducted with study participants for 4 weeks. One evening per week.
  Interventions: Behavioral: Mindfulness-based Stress Resilience Training
- Active Control Intervention (Active Comparator): Health Enhancement Program: This is a validated active comparator used in Mindfulness-based training studies. It will be conducted with the participants one evening per week for 4 weeks.
  Interventions: Behavioral: Health Enhancement Program

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Resilience Training — Mindfulness is a form of cognitive training that cultivates self-regulative ability and enhances resilience
  Arms: Experimental Intervention
Behavioral: Health Enhancement Program — This is a validated active control developed to serve as a control for mindfulness-based studies.
  Arms: Active Control Intervention

SUMMARY:
The objective of this study is to understand the prevalence of adverse childhood experiences (ACE) in students and to determine whether Mindfulness based stress resilience training (MBSR) is effective for promoting mental health in students with high ACE scores (>3). A double-blind randomized control study will examine the efficacy of MBSR in promoting positive change in measures of hope, rumination, forgiveness and stress.

DETAILED DESCRIPTION:
The Adverse Childhood Experiences Study examined the physical health and psychosocial consequences of ACE across the lifespan. This study demonstrated adverse childhood experiences (ACE) prevalence to be high and a direct correlation between ACE scores (a tally of different types of abuse, neglect, and household dysfunction experienced under the age of 18) and prevalence of physical health and psychosocial problems in adulthood. Adults with >3 ACE are more likely to experience social underachievement (e.g. lower educational achievement and economic productivity), physical and mental health problems (e.g. depression, heart disease, suicide attempts, substance abuse) and unhealthy lifestyle behaviours (e.g. smoking, physical inactivity). Worldwide, ACE have been shown to be prevalent, independent of social and economic factors, and highly interrelated. 12.5% of subjects reported >4 ACE. Among post-secondary students, studies determined high ACE scores to be associated with higher prevalence of risk behaviours and physical health and psychosocial problems. Failure to support the physical and mental health of students can lead to increased attrition, deterioration of well-being, and intentional self-harm.

Recognition of ACE prevalence and its consequences has been paralleled by the development of interventions for mitigating the lifetime health and social consequences of ACE. A 2016 study examining interventions believed to improve the mental health of adults with significant ACE (>3) identified mindfulness-based therapies (MBT) as being effective. Mindfulness is a form of cognitive training that cultivates self-regulative ability and enhances resilience.

As no Canadian post-secondary institution has comprehensively investigated the prevalence of student ACE, the objective of this study is to understand the prevalence of ACE in students and to determine whether MBT is effective for promoting mental health in students with high ACE scores (>3).

A double-blind randomized control study will examine the efficacy of MBT, specifically Mindfulness-based Stress Resilience Training (MBSR), in promoting positive change in measures of hope, rumination, forgiveness and distress. Interventions that positively effect these measures are known to enhance quality of life. First year students enrolled at Dalhousie University will be recruited. Subjects will complete an ACE questionnaire and those with >3 ACE prior to age 18 will be invited to participate in this study. Students with prior MBT training will be excluded. Subjects will be randomized to one of two groups: MBSR or an established active control (Health Enhancement Program (HEP)). We selected MBSR because it is secular, codified, and the most scientifically studied mindfulness-based intervention to date. Power analyses determined 25 subjects per group is sufficient to detect a significant difference in outcomes across the groups. Interventionists and subjects will be blinded. Students will be led in group based MBSR or HEP for 4 weeks. Prior to and after the 4-week intervention subjects' outcomes will be determined using the: Perceived Stress Scale; Rumination and Reflection Questionnaire; Heartland Forgiveness Scale and; Adult Dispositional Hope Scale.

Development of evidence-based programs that support the identification of ACE in students and identification of interventions that mitigate negative lifetime consequences of ACE outcomes is needed. This pilot study will increase understanding of Canadian student ACE and assess the effectiveness of MBSR as a tool for supporting the mental health of students who have experienced significant ACE.

ELIGIBILITY:
Inclusion Criteria:

* Post-secondary education students who are over the age of 18 and who had experienced more than 3 Adverse Childhood Experiences

Exclusion Criteria:

* Persons who had received prior training in mindfulness based approaches.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Stress | Pre and Post intervention (1 week)
  Measure of current stress using the Perceived Stress Scale
Rumination and Reflection | Pre and post intervention (1 week)
  Measured using the Rumination and Reflection Questionnaire
Forgiveness | Pre and post intervention (1 week)
  Measures using the Heartland Forgiveness Scale
Hope | Pre and post intervention (1 week)
  Measured using the Adult Dispositional Hope Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ross, PhD, Study Director — School of Social Work, Faculty of Health,Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No